CLINICAL TRIAL: NCT03742245
Title: Multicenter Phase I/Ib Trial of Olaparib in Combination With Vorinostat in Patients With Relapsed/Refractory and/or Metastatic Breast Cancer
Brief Title: Olaparib in Combination With Vorinostat in Patients With Relapsed/Refractory and/or Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: AstraZeneca (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Polly A. Niravath, MD, Section Chief, Breast Oncology, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00020138
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer Metastatic; Breast Cancer
Keywords: breast cancer; relapsed; refractory; metastatic
MeSH Terms: conditions — Breast Neoplasms; Recurrence; Neoplasm Metastasis | interventions — olaparib; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Olaparib and Vorinostat (Experimental): Phase I: Olaparib and vorinostat will be orally administered for 4 28-day cycles. Dose levels (DLs) are as follows: DL -1, 100 mg twice daily (b.i.d.) olaparib and 300 mg for 5 consecutive days per week vorinostat; DL 0 (starting dose), 200 mg twice daily (b.i.d.) olaparib and 300 mg once daily (q.d.) vorinostat; DL 1, 300 mg b.i.d. olaparib and 300 mg q.d. vorinostat; and DL 2, 300 mg b.i.d. olaparib and 400 mg q.d. vorinostat. . Patients who derive clinical benefit (CR, PR, or SD) after 4 cycles of treatment can continue to receive the study treatment until they experience unacceptable AEs or disease progression.
  Phase Ib: Olaparib and vorinostat will be administered at the maximum tolerated dose (MTD) determined in the Phase I portion of the study for 4 28-day cycles. Participants who derive clinical benefit (complete response, partial response, or stable disease) after 4 cycles will continue to receive study treatment until unacceptable toxicity or disease progression.
  Interventions: Drug: Olaparib; Drug: Vorinostat

INTERVENTIONS:
Drug: Olaparib — PARP inhibitor
  Other Names: AZD2281; KU-0059436; Lynparza
Drug: Vorinostat — HDAC inhibitor
  Other Names: Suberanilohydroxamic acid; Zolinza

SUMMARY:
The purpose of this study is to test the safety and preliminary efficacy of olaparib and vorinostat when used together in participants with relapsed/refractory and or metastatic breast cancer.

DETAILED DESCRIPTION:
This is a Phase I/Ib study testing the safety and preliminary efficacy of olaparib and vorinostat when used together in participants with relapsed/refractory and or metastatic breast cancer. Cancer cells grow in an uncontrolled manner and this causes damage to their DNA (genetic makeup). Cancer cells that cannot repair this damage will not survive and die. Unfortunately, cancer cells contain certain proteins whose job is to repair DNA damage. Poly (adenosine 5' diphosphoribose) polymerase (PARP) and histone deacetylase (HDAC) are two such proteins. Olaparib stops PARP from working, and vorinostat stops histone deacetylase from working. The use of olaparib and vorinostat together may better block the ability of cancer cells to repair their DNA damage. This may lead to even better killing of cancer cells.

The study will be done in two parts. In part one of the study, different dose levels of olaparib and vorinostat will be tested in several study participants. This part of the study will allow us to see the doses of olaparib and vorinostat that can be used safely together in participants with relapsed/refractory and/or metastatic breast cancer. Up to 4 different dose levels will be studied. In part two of the study, the dose level of olaparib and vorinostat found to be the safest in the first part of the study will be tested. This part of the study will allow us to see how well relapsed/refractory and/or metastatic breast cancer responds to treatment with olaparib and vorinostat. Participants who received the dose level of olaparib and vorinostat found to be the safest in the first part of the study will also take part in part two of the study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study-specific procedures.
* Female or male ≥18 years of age.
* Histologically or cytologically confirmed relapsed/refractory and/or metastatic breast cancer with the exception of human epidermal growth factor receptor 2-positive breast cancer.
* Evaluable or measurable disease as per the RECIST 1:1.
* Normal organ and bone marrow function measured within 28 days prior to administration of the study treatment.
* White blood cell (WBC) count >2,500/microL and <15,000/microL
* Lymphocyte count ≥500/microL
* Total bilirubin (TBL) ≤1.5 × institutional ULN
* Serum aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤2.5 × institutional ULN (patients with liver metastases ≤5 × ULN) and alkaline phosphatase (ALP) ≤2.5 × institutional ULN (patients with liver metastases ≤5 × ULN).
* Serum creatinine ≤1.5 × ULN and creatinine clearance (CrCl) estimated using the Cockcroft-Gault equation of ≥51 mL/min
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* Life expectancy ≥6 months.
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential (WOCBP): negative serum (beta-human chorionic gonadotropin) pregnancy test within 28 days of study treatment and confirmed prior to treatment on Day 1.
* WOCBP must be willing to use 2 highly effective methods of contraception for the course of the study through 1 month after the last treatment dose.
* Male patients must be willing to use condom contraception for the course of the study through 3 months after the last treatment dose.
* Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
* Willing to undergo biopsy as required by the study.
* Able to swallow pills and capsules

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation.
* Whole blood transfusions in the last 120 days prior to study entry.
* Unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study treatment.
* Concomitant use of known strong or moderate cytochrome P450 (CYP)3A inhibitors.
* Concomitant use of known strong or moderate CYP3A inducers.
* Persistent toxicities (CTCAE Grade 2) caused by previous cancer therapy, excluding alopecia.
* Participants with myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with features suggestive of MDS/AML.
* Known hypersensitivity to olaparib or vorinostat or any of their excipients or analogues (PARP/HDAC inhibitors).
* Breastfeeding women.
* No active malignancy except for non-melanoma skin cancer, in situ cervical cancer, or a treated cancer from which the patient has been continuously disease free for more than 5 years.
* Pneumonitis or at risk of pneumonitis.
* Uncontrolled brain or leptomeningeal metastases.
* Any systemic chemotherapy or radiation therapy within 4 weeks prior to study entry.
* Major surgery within 4 weeks of starting the study treatment.
* Participation in another clinical study with an investigational product during the last 3 months.
* Any previous treatment with PARP inhibitor including olaparib or HDAC inhibitor including vorinostat.
* New York Heart Association Class III or IV heart failure or unstable angina.
* History of liver disease, such as cirrhosis or active/chronic hepatitis B or C.
* Sustained or clinically significant cardiac arrhythmias including sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, advanced heart block (Mobitz II or higher atrioventricular nodal block), prolonged corrected QT interval (mean >470 milliseconds), or history of acute myocardial infarction.
* Risk factors for torsades de pointes such as hypokalemia, hypomagnesemia, cardiac failure, clinically significant/symptomatic bradycardia, or high-grade atrioventricular nodal block.
* Concomitant disease(s) that could prolong QT interval such as autonomic neuropathy (caused by diabetes or Parkinson's disease), human immunodeficiency virus (HIV), cirrhosis, uncontrolled hypothyroidism, or cardiac failure.
* Concomitant medication(s) known to prolong QT interval (patient must be off the drug for 2 weeks to be eligible).
* Presence of active or suspected acute or chronic uncontrolled infection or history of immunocompromise, including participants who are known to be serologically positive for HIV.
* Any severe and/or uncontrolled medical conditions or other conditions that could affect study participation, such as severely impaired lung function; any active (acute or chronic) or uncontrolled infection/disorders; or non-malignant medical illnesses that are uncontrolled or whose control may be jeopardized by the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-06-11 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
MTD | 16 weeks
  Determine the MTD of the olaparib and vorinostat combination

SECONDARY OUTCOMES:
Dose-limiting toxicities (DLTs) and other adverse events | 16 weeks
  Determine the DLTs and other adverse events associated with the olaparib and vorinostat combination, as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v4.03
Recommended Phase 2 dose (RP2D) | 16 weeks
  Determine the RP2D of the olaparib and vorinostat combination
Antitumor activity | 16 weeks
  Assess the antitumor activity of the olaparib and vorinostat combination in an expansion cohort of patients with relapsed/refractory and/or metastatic breast cancer, as assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) 1:1

CONTACTS AND LOCATIONS:
Overall Officials: Polly Niravath, M.D., Principal Investigator — Houston Methodist Cancer Center
Locations (1):
- Houston Methodist Cancer Center, Houston, Texas, United States